CLINICAL TRIAL: NCT03852316
Title: Pivotal Study of a Single-Use, Point-of-Care Molecular Diagnostic Device for the Detection of Neisseria Gonorrhoeae (NG), Trichomonas Vaginalis (TV), and Chlamydia Trachomatis (CT) in Women
Brief Title: Clinical Study of a Diagnostic Device for NG, TV and CT in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0024
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2019-02

CONDITIONS: Chlamydial Infection; Gonococcal Infection; Trichomoniasis
Keywords: Chlamydia trachomatis; Device; Diagnostic; Neisseria gonorrohoeae; Trichomonas vaginalis
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Trichomonas Infections; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Click Device (Experimental): Each subject (females 14 years of age and older) will perform a self-collection vaginal swab for the Click device and be randomized to a particular order for three vaginal swab collections (performed by Health Care Providers (HCP) as defined by state/local regulatory authorities) for comparator methods. N=1750
  Interventions: Device: Click Device

INTERVENTIONS:
Device: Click Device — A single-use device containing a polymerase chain reaction (PCR)-based nucleic acid amplification test (NAAT) for detection of deoxyribonucleic acid (DNA) from Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Trichomonas vaginalis (TV) in self-collected vaginal specimens.

SUMMARY:
This is a multi-center study with a minimum of three sites in the United States. The study will enroll approximately 1750 female subjects, 14 years of age and older, and will have a study duration of approximately 9 months after enrollment of the first subject. Female subjects seen at the participating sites for any reason will be evaluated for enrollment in this study. All subjects will be managed per standard of care as applicable. Subjects who are enrolled in the study will perform self-collection of a vaginal swab to be tested by Click device and allow the health care provider (HCP) to collect three additional vaginal swabs to be tested by recognized FDA-cleared comparator methods. Subjects will complete the study in a single visit. The primary objective is to assess the performance of the Click device for detection of Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Trichomonas vaginalis (TV) in self-collected vaginal specimens as compared to Patient Infected Status (PIS) determined by three approved comparator assays using vaginal specimens collected by a qualified HCP in support of obtaining FDA clearance. and a Clinical Laboratory Improvement Amendments (CLIA) Waiver.

DETAILED DESCRIPTION:
This is a multi-center study with a minimum of three clinical sites across diverse geographical areas in the United States. Approximately one-third of the total number of sites will have a patient population of low Neisseria gonorrhoeae (NG), Chlamydia trachomatis (CT), or Trichomonas vaginalis (TV) prevalence. Low prevalence sites are defined as sites with a prevalence < / = 2 percent for any of the three targets. Sites with a prevalence higher than 2 percent for any of the three targets will be defined as high prevalence sites. The study will enroll approximately 1750 female subjects, 14 years of age and older, and will have a study duration of approximately 9 months after enrollment of the first subject. Female subjects seen at the participating sites for any reason will be evaluated for enrollment in this study. All subjects will be managed per standard of care as applicable. Subjects who are enrolled in the study will perform self-collection of a vaginal swab to be tested by Click device and allow the health care provider (HCP) to collect three additional vaginal swabs to be tested by recognized FDA-cleared comparator methods. Subjects will complete the study in a single visit, approximately 60 minutes in length. The hypothesis of this study is that Click Diagnostics Sexual Health Test performs substantially equivalent to the NAAT (Nucleic Acid Amplification Test) predicate system, and the identification of each organism (CT, NG, and TV) in self-collected vaginal swabs by women using the Click device will agree with the Patient Infected Status (PIS) with a high sensitivity and specificity. The primary objective is to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP in support of obtaining FDA clearance and a Clinical Laboratory Improvement Amendments (CLIA) Waiver. The secondary objectives are: 1) to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens among symptomatic subjects as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP; 2) to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens among asymptomatic subjects as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give voluntary written informed consent (or the parent/legal guardian will provide parental permission) before any study-related procedure is performed.
2. Female at birth. (Pregnant and breastfeeding women are eligible.)
3. Age > / = 14 years at the time of enrollment.
4. Able to read and understand the procedural information provided for the study.
5. Able and willing to follow all study procedures, including performing self-collection of one vaginal swab and permitting a licensed HCP to collect three additional vaginal swabs.

Exclusion Criteria:

1. Have a medical condition, serious intercurrent illness, or other circumstance that, in the Investigator's judgment, could jeopardize the subject's safety, or could interfere with study procedures.
2. Enrollment in this study previously.
3. Use of antiperspirants and deodorants or the following vaginal products: douches, washes, lubricants, vaginal wipes, vaginal moisturizers, or feminine hygiene spray in the genital area, within 48 hours prior to enrollment.

Ages: 14 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1585 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Axis Clinical Trials, Los Angeles, California
  - University of California, San Diego - Antiviral Research Center, San Diego, California
  - San Francisco Department of Public Health - San Francisco City Clinic, San Francisco, California
  - South Florida Clinical Trials, Hialeah, Florida
  - Florida International University - Student Health Center, Miami, Florida
  - Cook County Health and Hospitals System - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - University of Mississippi - Infectious Diseases, Jackson, Mississippi
  - Impact Clinical Trials, Las Vegas, Nevada
  - Philadelphia Department of Public Health - Health Center 1, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were females 14 to 80 years of age, inclusive, recruited from 10 clinic sites across 7 states at locations including but not limited to: OB/GYN and primary care offices, as well as sexually transmitted disease, teen, public health, and family planning clinics. Participants were enrolled from 27FEB2019 to 02DEC2019.
Groups:
- Click Device: Female participants >=14 years of age who may have been symptomatic or asymptomatic for sexually transmitted infections (STIs). Participants who met the inclusion/exclusion criteria and were enrolled performed self-collection with a vaginal swab for the Click device, and allowed the health care professional (HCP) to collect three additional vaginal swabs for the comparator methods.
Period: Overall Study
Arm/Group | Click Device
Started | 1585
Completed | 1581
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Enrolled but Device not Utilized | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants that were enrolled in the study.
Groups:
- Click Device: Female participants >=14 years of age who may have been symptomatic or asymptomatic for STIs. Participants who met the inclusion/exclusion criteria and were enrolled performed self-collection with a vaginal swab for the Click device, and allowed the health care professional (HCP) to collect three additional vaginal swabs for the comparator methods.
Arm/Group | Click Device
Number analyzed (Participants) | 1585
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1551
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1585
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 310
  Not Hispanic or Latino | 1168
  Unknown or Not Reported | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12
  Asian | 86
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 876
  White | 414
  More than one race | 70
  Unknown or Not Reported | 121
Region of Enrollment [Number; unit: participants]
  United States | 1585
Evaluable Results [Count of Participants; unit: Participants] — This population includes participants with a valid Click and valid PIS result for the pathogen in question.
  Participants
    C.trachomatis | 1457
    N. gonorrhoeae | 1468
    T. vaginalis | 1449
Symptomatic Status [Number; unit: participants] — Population: The number analyzed represents the number of participants that reported a valid Click and a valid PIS result for the pathogen in question.
  participants
    C. trachomatis : Symptomatic: number analyzed (Participants) | 1457
    C. trachomatis : Symptomatic | 735
    C. trachomatis : Asymptomatic: number analyzed (Participants) | 1457
    C. trachomatis : Asymptomatic | 722
    N. gonorrhoeae : Symptomatic: number analyzed (Participants) | 1468
    N. gonorrhoeae : Symptomatic | 746
    N. gonorrhoeae : Asymptomatic: number analyzed (Participants) | 1468
    N. gonorrhoeae : Asymptomatic | 722
    T. vaginalis : Symptomatic: number analyzed (Participants) | 1449
    T. vaginalis : Symptomatic | 734
    T. vaginalis : Asymptomatic: number analyzed (Participants) | 1449
    T. vaginalis : Asymptomatic | 715

OUTCOME MEASURES:

1. Primary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device for Detection of Chlamydia Trachomatis (CT) in Self-collected Vaginal Specimens as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP
Description: The sensitivity of the Click device is defined as follows:
  TP = the number of specimens where both the Click result and the PIS designation are Positive.
  FN = the number of specimens where the Click result is Negative and the PIS designation is Positive.
  Sensitivity = 100 * TP / (TP + FN)
  The specificity of the Click device is defined as follows:
  TN = the number of specimens where both the Click result and the PIS designation are Negative.
  FP = the number of specimens where the Click result is Positive and the PIS designation is Negative.
  Specificity = 100 * TN / (TN + FP)
Time Frame: Day 1
Population: Evaluable Population: This population included all samples which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 1457
percentage of participants
  Sensitivity | 97.6 [93.2 to 99.2]
  Specificity | 98.3 [97.5 to 98.9]

2. Primary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device for Detection of Neisseria Gonorrhoeae (NG) in Self-collected Vaginal Specimens as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP
Description: as for outcome 1
Time Frame: Day 1
Population: Evaluable Population: This population included all samples which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 1468
percentage of participants
  Sensitivity | 97.4 [86.5 to 99.5]
  Specificity | 99.4 [98.9 to 99.7]

3. Primary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device for Detection of Trichomonas Vaginalis (TV) in Self-collected Vaginal Specimens as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP
Description: as for outcome 1
Time Frame: Day 1
Population: Evaluable Population: This population included all samples which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 1449
percentage of participants
  Sensitivity | 99.2 [95.5 to 99.9]
  Specificity | 96.9 [95.8 to 97.7]

4. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of CT From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Asymptomatic Participants
Description: If a participant reported "Yes" to any of the following symptoms, the participant is classified as Symptomatic: Unusual vaginal discharge; Vaginal irritation (itching, burning, soreness); Lower abdominal/pelvic pain; Painful urination; Increased urinary frequency; Abnormal bleeding/spotting; Pain or bleeding with sex/intercourse. Otherwise, the participant is classified as "Asymptomatic".
  The sensitivity of the Click device is defined as follows:
  TP = the number of specimens where both the Click result and the PIS designation are Positive.
  FN = the number of specimens where the Click result is Negative and the PIS designation is Positive.
  Sensitivity = 100 * TP / (TP + FN)
  The specificity of the Click device is defined as follows:
  TN = the number of specimens where both the Click result and the PIS designation are Negative.
  FP = the number of specimens where the Click result is Positive and the PIS designation is Negative.
  Specificity = 100 * TN / (TN + FP)
Time Frame: Day 1
Population: Evaluable Asymptomatic Population: This population included all samples from asymptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 722
percentage of participants
  Sensitivity | 95.8 [86.0 to 98.8]
  Specificity | 99.0 [97.9 to 99.5]

5. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of NG From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Asymptomatic Participants
Description: as for outcome 4
Time Frame: Day 1
Population: Evaluable Asymptomatic Population: This population included all samples from asymptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 722
percentage of participants
  Sensitivity | 94.4 [74.2 to 99.0]
  Specificity | 99.4 [98.5 to 99.8]

6. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of TV From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Asymptomatic Participants
Description: as for outcome 4
Time Frame: Day 1
Population: Evaluable Asymptomatic Population: This population included all samples from asymptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 715
percentage of participants
  Sensitivity | 100 [92.7 to 100]
  Specificity | 98.0 [96.7 to 98.9]

7. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of CT From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 4
Time Frame: Day 1
Population: Evaluable Symptomatic Population: This population included all samples from symptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 735
percentage of participants
  Sensitivity | 98.7 [93.0 to 99.8]
  Specificity | 97.7 [96.3 to 98.6]

8. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of NG From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 4
Time Frame: Day 1
Population: Evaluable Symptomatic Population: This population included all samples from symptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 746
percentage of participants
  Sensitivity | 100 [83.9 to 100]
  Specificity | 99.4 [98.6 to 99.8]

9. Secondary Outcome: The i) Percent Sensitivity and ii) Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of TV From Self-collected Specimens as Compared to PIS Using Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 4
Time Frame: Day 1
Population: Evaluable Symptomatic Population: This population included all samples from symptomatic participants which provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. A sample provides an evaluable result if both the Click device and the PIS provide a valid positive or negative result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Click Device
Number analyzed (Participants) | 734
percentage of participants
  Sensitivity | 98.6 [92.6 to 99.8]
  Specificity | 95.8 [93.9 to 97.1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the time of swab collection to the time that the participant left the clinic on the same day.
Arm/Group | Click Device
All-Cause Mortality (participants affected / at risk) | 0/1585
Serious Adverse Events (participants affected / at risk) | 0/1585
Other Adverse Events (participants affected / at risk) | 0/1585

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03852316/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03852316/SAP_002.pdf
  • Informed Consent Form (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03852316/ICF_000.pdf